CLINICAL TRIAL: NCT00606151
Title: Short-Term Outcomes of Perioperative Anticoagulation in the Setting of Recent Intracoronary Drug Eluting Stents
Brief Title: PeriOperative Bridging - Perioperative Anticoagulation in the Setting of Recent Intracoronary Drug Eluting Stents
Status: Terminated | Type: Observational
Why Stopped: subject enrollment goals not met
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Matthew Becker, MD, Cleveland Clinic
Other Study IDs: 07669; 07669
Record Dates: First submitted 2008-01-22; First posted 2008-02-01 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Stent Thrombosis
Keywords: drug eluding stents; perioperative bridging; Stents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if an intravenous (IV) antiplatelet medication is as safe and effective at preventing clot formation in your stented artery as compared in people who have stopped clopidogrel prior to surgery.

DETAILED DESCRIPTION:
Stent thrombosis continues to be associated with a high rate of death or myocardial infarction. While this risk has been ameliorated through the use of the oral antiplatelet agent clopidogrel, there is a small but important subset of patients who will require discontinuation of clopidogrel due to unplanned or emergency surgery. These patients are exposed to a high risk of stent thrombosis during this time period. It is not known whether a strategy of intravenous antiplatelet therapy to "bridge" these patients is effective at preventing the morbidity related to stent thrombosis in the perioperative period. We intend to assess, in a prospective observational manner, the clinical course of patients who have undergone stent implantation less than 6 months prior to a surgical procedure requiring discontinuation of clopidogrel therapy and the efficacy of intravenous antiplatelet therapy to prevent morbidity related to stent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or greater, able to give consent
* DES implantation < or = 6 months prior to admission
* Undergoing an invasive surgical procedure that will require cessation of clopidogrel therapy for >48 hours

Exclusion Criteria:

* Age < 18 years
* Refusal to give consent
* Surgical procedure performed without discontinuation of clopidogrel therapy (or < 48h of clopidogrel cessation)
* Ongoing anticoagulant therapy other than aspirin (i.e. warfarin, ticlopidine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We intend to assess, in a prospective observational manner, the clinical course of patients who have undergone stent implantation less than 6 months prior to a surgical procedure requiring discontinuation of clopidogrel therapy and the efficacy of intravenous antiplatelet therapy to prevent morbidity related to stent thrombosis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
stent thrombosis | hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Matthew (Casey) Becker, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States